CLINICAL TRIAL: NCT02209025
Title: The Effects of Short-term Theobromine Supplementation on Vascular Function and Intestinal apoA-I Production in Fasting and in the Postprandial State
Brief Title: Theobromine, Vascular Function and Intestinal apoA-I Production
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Unilever R&D (Industry); DSM Nutritional Products, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NL46131.068.13/METC 13-3-065
Record Dates: First submitted 2014-08-04; First posted 2014-08-05 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2014-08

CONDITIONS: Cardiovascular Disease
Keywords: Atherosclerosis; Cholesterol; Cholesterol, HDL; Apolipoprotein A-I; Theobromine
MeSH Terms: conditions — Cardiovascular Diseases; Atherosclerosis | interventions — Theobromine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo drink (Placebo Comparator): A drink with the same components as the theobromine drink except for the theobromine
  Interventions: Dietary Supplement: Placebo drink
- Theobromine (Experimental): 500mg theobromine in a drink
  Interventions: Dietary Supplement: Theobromine

INTERVENTIONS:
Dietary Supplement: Theobromine — Theobromine a compound for cocoa
  Arms: Theobromine
Dietary Supplement: Placebo drink
  Arms: Placebo drink

SUMMARY:
Rationale: Despite successful efforts to lower atherogenic serum low-density lipoprotein (LDL) cholesterol concentrations, a substantial residual cardiovascular risk remains. An additive strategy to further lower this residual risk may be via raising high-density lipoprotein (HDL) concentrations, and in particular those of its major protein constituent apolipoprotein A-I (apoA-I). Based on several studies, theobromine may be a promising candidate in this respect. Recently, theobromine was shown to increase serum HDL cholesterol (HDL-C) concentrations by 0.16 mmol/L or 10% and apoA-I levels with 8%. The question is whether this increase in HDL-C and apoA-I concentrations observed translates into an improved functionality of the blood vessels. Effects of theobromine on vascular function have never been evaluated in a placebo controlled human intervention study.

Objective: The primary objective is to evaluate the long-term effects of theobromine on vascular function in healthy subjects with a slightly lowered HDL-C in the fasting and the postprandial state. The second primary objective is to evaluate the long-term effects of theobromine on intestinal apoA-I mRNA and protein expression levels in healthy subjects with a slightly lowered HDL-C in the fasting and the postprandial state.

Secondary objectives are to study the long-term effects of theobromine on (1) fasting serum HDL-C concentrations, (2) cholesterol efflux capacity and (3) postprandial lipid and glucose metabolism.

Study design: A randomized, double-blind, placebo controlled cross-over design. The total study duration will be 12 weeks, consisting of a 4 week experimental period, a 4 week wash-out, and a 4 week control period. At the end of the experimental and control periods, a postprandial test will take place.

Study population: Forty-eight healthy men aged 45-70 years and women aged 50-70 years, with slightly lowered HDL-C concentrations (men <1.3 mmol/L and women <1.5 mmol/L).

Intervention: During the experimental period, subjects will consume daily at breakfast an drink containing 500 mg theobromine. During the placebo period, the subjects will consume daily at breakfast the same drink without theobromine. During the wash-out period, they will not consume any of the drinks.

Main study parameters/endpoints: Measurements will be performed at the end of both 4-week intervention periods. The effects of theobromine will be calculated as the absolute differences between values obtained at the end of each period. The primary endpoint is the change in vascular function defined as % change in flow-mediated dilation (FMD) after intake of a daily stressor, a milkshake providing all the three different macronutrients. The second primary endpoint is the change in apoA-I mRNA and protein expression on the end of each period 5 hours after intake of the milkshake.

DETAILED DESCRIPTION:
Rationale: Despite successful efforts to lower atherogenic serum low-density lipoprotein (LDL) cholesterol concentrations, a substantial residual cardiovascular risk remains. An additive strategy to further lower this residual risk may be via raising high-density lipoprotein (HDL) concentrations, and in particular those of its major protein constituent apolipoprotein A-I (apoA-I). Based on several studies, theobromine may be a promising candidate in this respect. Recently, theobromine was shown to increase serum HDL cholesterol (HDL-C) concentrations by 0.16 mmol/L or 10% and apoA-I levels with 8%. The question is whether this increase in HDL-C and apoA-I concentrations observed translates into an improved functionality of the blood vessels. Effects of theobromine on vascular function have never been evaluated in a placebo controlled human intervention study.

Objective: The primary objective is to evaluate the long-term effects of theobromine on vascular function in healthy subjects with a slightly lowered HDL-C in the fasting and the postprandial state. The second primary objective is to evaluate the long-term effects of theobromine on intestinal apoA-I mRNA and protein expression levels in healthy subjects with a slightly lowered HDL-C in the fasting and the postprandial state.

Secondary objectives are to study the long-term effects of theobromine on (1) fasting serum HDL-C concentrations, (2) cholesterol efflux capacity and (3) postprandial lipid and glucose metabolism.

Study design: A randomized, double-blind, placebo controlled cross-over design. The total study duration will be 12 weeks, consisting of a 4 week experimental period, a 4 week wash-out, and a 4 week control period. At the end of the experimental and control periods, a postprandial test will take place.

Study population: Forty-eight healthy men aged 45-70 years and women aged 50-70 years, with slightly lowered HDL-C concentrations (men <1.3 mmol/L and women <1.5 mmol/L).

Intervention: During the experimental period, subjects will consume daily at breakfast an drink containing 500 mg theobromine. During the placebo period, the subjects will consume daily at breakfast the same drink without theobromine. During the wash-out period, they will not consume any of the drinks.

Main study parameters/endpoints: Measurements will be performed at the end of both 4-week intervention periods. The effects of theobromine will be calculated as the absolute differences between values obtained at the end of each period. The primary endpoint is the change in vascular function defined as % change in flow-mediated dilation (FMD) after intake of a daily stressor, a milkshake providing all the three different macronutrients. The second primary endpoint is the change in apoA-I mRNA and protein expression on the end of each period 5 hours after intake of the milkshake.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Before the study, subjects will be screened twice to determine eligibility during two visits of 15 minutes. During these visits, body weight, height and blood pressure will be measured. In addition, a venous blood sample (5.5 mL at each occasion) will be drawn. During the study, subjects will receive the control and theobromine drinks in random order. At day 1 and 14 a fasting venous blood sample (16.5 mL and 7 mL respectively) will be drawn and body weight and blood pressure will be measured. At days 25 and 81 again a fasting blood sample will be drawn (28 mL). In addition, at day 28 of each experimental period, at t=0 hours, a fasting venous blood sample (30 mL) will be drawn and vascular function will be measured, followed by a 2.5 h postprandial test with again the vascular function measurements. As postprandial meal, subjects will receive a high-fat milkshake. Before the postprandial test a cannula will be placed and blood will be sampled at t=0, 15, 30, 45, 60, 90, 120 and 240 (total volume 129.5 mL). Thus, during the entire 13 (screening and study) weeks period, in total 444 mL blood will be drawn. Vascular function measurements include a panel of non-invasive measurements, i.e. FMD, endo peripheral artherial tonometry (endoPAT), pulse wave velocity (PWV) and retinal imaging. Subjects will be asked to fill out a food frequency questionnaire two times and to keep a study-diary throughout 12 weeks. On rare occasions, blood sampling might cause bruises or hematoma. The vascular function measurements are non-invasive and will cause no burden.

In a subgroup of 10 volunteers, 5 hours after the start of the postprandial test, small intestinal biopsies will be taken in the duodenum to determine the difference in intestinal apoA-I mRNA and protein expression. Obtaining small intestinal biopsies by standard flexible gastroscopy induces local discomfort in the pharynx only during the procedure, which takes about 15 minutes, and causes a theoretical risk for perforations (1:1000) and an infection risk of 1:1.800.000, with lower risk for healthy subjects. The complication is serious and subjects will have to stay in the hospital. If there are serious complaints after the gastroscopy (e.g. vomiting with or without blood, or stomach ache) subjects are have to warn the project leader or their physician.

Total time investment for the subjects will be approximately 14.5 hours, and 17.5 hours in the subgroup from which biopsies will be taken, excluding travel time.

ELIGIBILITY:
Inclusion Criteria:

* Men aged between 45 and 70 years,
* Women aged between 50 and 70 years,
* Serum HDL-C <1.3 mmol/L (men),
* Serum HDL-C <1.5 mmol/L (women),
* Serum total cholesterol <8.0 mmol/L,
* Plasma glucose <7.0 mmol/L,
* BMI between 25 - 35 kg/m2,
* Non-smoking,

Exclusion Criteria:

* Unstable body weight (weight gain or loss >3 kg in the past 3 months),
* Any medical condition requiring treatment and/or medication use,
* Indication for treatment with cholesterol-lowering drugs according to the Dutch Cholesterol Consensus (30),
* Use of medication or a medically-prescribed diet known to affect serum lipid or glucose metabolism. The use of paracetamol is allowed.
* Active cardiovascular disease (for instance congestive heart failure) or recent (<6 months) event, such as acute myocardial infarction or cerebro-vascular accident.
* Gastrointestinal diseases (like celiac disease, inflammatory bowel disease, irritable bowel disease and food allergies) or a history of any gastrointestinal disorders or complaints.
* Not willing to stop the consumption of vitamin supplements or fish oil capsules 2 weeks before the start of the study,
* Men: consumption of >21 glasses of alcohol-containing drinks per week.
* Women: consumption of >14 glasses of alcohol-containing drinks per week.
* Abuse of drugs,
* Extensive exercise,
* Not willing to abstain from caffeine containing painkillers two weeks prior to the study and the duration of the study,
* Not willing to abstain from theobromine rich products from two weeks prior to the study and the duration of the study:

  o Chocolate containing products (see Appendix A).
* Not willing to abstain from energy drinks from two weeks prior to the study and the duration of the study, because of the high caffeine content.
* Not willing to reduce caffeine containing drinks till maximum 4 drinks a day from two weeks prior to the study and the duration of the study:

  * Coffee (excluding coffee without caffeine) (see Appendix A),
  * Tea (excluding tea without caffeine) (see Appendix A),
  * Cola (see Appendix A).
* Participation in another biomedical study within 1 month prior to the screening visit,
* Having donated >150 ml blood within 1 month prior to the screening visit, planning to donate blood during the study or within one month after finishing the study.
* Impossible or difficult to puncture as evidenced during the screening visits.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-06; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Flow mediated dilation | 4 weeks
  FMD measurements after 4 weeks of intake. Fasting and postprandial measurements
Intestinal apoA-I production | After 4 weeks of intake
  Intestinal biopsies after 4 weeks of intake to see changes in apoA-I gene expression

SECONDARY OUTCOMES:
HDL cholesterol | 4 weeks
  HDL serum cholesterol concentrations after 4 weeks of intake
Vascular measurements | After 4 weeks
  Vascular function measurements (PAT, PWV, PWA, retinal images) after 4 weeks of intake.
  Fasting and postprandial measurements
serum lipid metabolism | 4 weeks
  serum lipid metabolism (total cholesterol, LDL-cholesterol, triglycerides) during fasting and in the postprandial state?
glucose metabolism | 4 weeks
  glucose and insulin concentrations during fasting and in the postprandial state?
(apo)lipoprotein metabolism | 4 weeks
  ApoB concentrations during fasting and in the postprandial state

CONTACTS AND LOCATIONS:
Overall Officials: J Plat, Prof, Principal Investigator — Maastricht University Hospital
Locations (1):
- Maastricht University Hospital, Maastricht, Netherlands

REFERENCES:
- [Derived] Smolders L, Mensink RP, van den Driessche JJ, Joris PJ, Plat J. Theobromine consumption does not improve fasting and postprandial vascular function in overweight and obese subjects. Eur J Nutr. 2019 Apr;58(3):981-987. doi: 10.1007/s00394-018-1612-6. Epub 2018 Jan 12. PMID 29330660
- [Derived] Smolders L, Mensink RP, Boekschoten MV, de Ridder RJJ, Plat J. Theobromine does not affect postprandial lipid metabolism and duodenal gene expression, but has unfavorable effects on postprandial glucose and insulin responses in humans. Clin Nutr. 2018 Apr;37(2):719-727. doi: 10.1016/j.clnu.2017.06.007. Epub 2017 Jun 10. PMID 28645636